CLINICAL TRIAL: NCT02914353
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate The Safety Tolerability, Pharmacokinetics, and Pharmacodynamcs of Single and Multiple Ascending Doses of EP-7041 in Hea;Thy Subjects
Brief Title: Study to Evaluate Safety, PK and PD of Single and Multiple Ascending Doses of EP-7041 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: eXIthera Pharmaceuticals (Industry)
Collaborators: IDT CMAX Clinical Trials (Unknown); Syneos Health (Other); CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXI-111
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Factor X!a; anticoagulant; thromboembolism; venous thromboembolism; embolism and thrombosis; enzyme inhibitors; hematologic agent
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism; Embolism and Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental - EP-7041 (Experimental): Single Ascending Dose: Single IV dose for each cohort; dose range 0.01 mg/kg to 1.0 mg/kg
  Multiple Ascending Dose: 0.01 mg/kg/h - 5 x 24 h continuous infusion up to 0.6 mg/kg/h - 5 x 24 h continuous infusion
  Interventions: Drug: EP=7041
- Placebo - Sterile Saline (Placebo Comparator): Single Ascending Dose: Single IV dose for each cohort;
  Multiple Ascending Dose: 5 x 24 h continuous infusion for each cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP=7041 — Factor X!a Inhibitor
  Arms: Experimental - EP-7041
Drug: Placebo — Normal Saline
  Arms: Placebo - Sterile Saline

SUMMARY:
This First-In-Human study will evaluate the safety and tolerability, pharmacokinetic profile, and pharmacodynamic effects of EP-7041, a novel Factor XIa inhibitor, following IV administration of single ascending doses in healthy normal volunteers, and following continuous IV infusions of multiple ascending doses in healthy normal volunteers.

DETAILED DESCRIPTION:
This will be a single-center, Phase 1a/1b, placebo-controlled, randomized, double-blind, integrated sequential ascending dose / multiple ascending dose study.

The study will be divided into two parts: the single ascending dose evaluation in healthy normal volunteers will constitute Part A and the multiple ascending doses evaluation in healthy normal volunteers will constitute Part B. The two study parts will be performed sequentially with partial overlapping.

Part A will include up to 6 cohorts (1 cohort per dose level; 4 planned cohorts and 2 optional adaptive cohorts). Each cohort will include 8 subjects - 6 on active drug and 2 on placebo - resulting in a maximum number of 48 subjects in the study - 32 planned and 16 optional. Subjects in each cohort will receive a single IV slow bolus (50 mL over 5 minutes) administration of study medication or placebo. The dose of EP-7041 will be sequentially escalated cohort by cohort in Part A . A staggered dosing schedule will be used for each cohort of Part A: 2 sentinel subjects (1 active and 1 placebo) will be dosed first and the remaining 6 subjects will be dosed the next day (5 active and 1 placebo).

Part B will include up to 4 cohorts (1 cohort per dose level; 3 planned cohorts and 1 optional adaptive cohort). As in Part A, each cohort of Part B will include 6 subjects on active drug and 2 on placebo, for a total of 8 subjects per cohort. Part B will therefore involve, at maximum, 32 subjects, with 24 planned subjects an 8 optional subjects. Subjects in each cohort of Part B will receive a total of 5 sequential 24-hour IV infusions of EP-7041 or matching placebo.

Evaluation of safety and tolerability to EP-7041 will include adverse events (i.e., seriousness, severity, relationship to EP-7041), vital signs, ECG, clinical laboratory parameters, physical examination, local response to each injection, and body weight.

Pharmacokinetic analyses will be performed with measurements of EP-7041 plasma concentrations, following single and multiple IV doses.

Pharmacodynamic effects of EP-7041 will be evaluated through the measurement of aPTT and PT in all subjects at multiple times throughout the course of both studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker (no use of tobacco products within 3 months prior to screening), ≥18 and ≤60 years of age, with Body Mass Index (BMI) > 18.5 and < 32.0 kg/m2 and a weight of at least 60 kg but not greater than 100 kg.
* Healthy as defined by:

  1. No history of abnormal bleeding episodes, e.g. nosebleeds, or abnormally heavy periods, or extensive bleeding after injury, surgery or dental work.
  2. A normal short physical examination and normal vital signs (heart rate (HR), blood pressure (BP) and tympanic body temperature).
  3. Normal laboratory tests (hematology, biochemistry, urinalysis, coagulation tests (aPTT and PT).
  4. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
  5. the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening which, at the investigator's discretion, warrants exclusion or positive test for hepatitis B, hepatitis C, or HIV.
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to drug administration.
* Positive pregnancy test at screening or check-in (Day -1).
* Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 160 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 40 or over 100 bpm) at screening or check-in (Day -1).
* Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics), or five (5) half-lives, whichever is longer, prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
* Hemoglobin or hematocrit clinically significantly less than lower limits of normal at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 following a single IV bolus of EP-7041 | Adverse events will be collected and documented during the course of the study. For a period of 30 days following the last study drug administration, adverse events will also be documented if reported.
  Assessment of safety and tolerability to EP-7041, administered as a single IV bolus, will be based on adverse events. Each AE will be graded with respect to its relationship to treatment using five categories: not related, unlikely, possible, probable, and highly probable. Each AE will also be graded on a three-point severity scale: mild, moderate, and severe. Adverse events will be coded by body system and preferred term using the MedDRA (Medical Dictionary for Regulatory Activities) dictionary. Assessments as to the effect of EP-7041 on vital signs, 12-lead ECG, telemetry, clinical laboratory parameters, physical examination, and local response to each injection, and body weight will also be made.
  The number and percentage of subjects experiencing adverse events will be tabulated for each treatment group by body system and preferred term. The number and percentage of subjects experiencing AEs will also be tabulated by relationship to drug treatment and by severity. If an AE is
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 following a continuous IV infusion of EP-7041 administered over 5 days | Adverse events will be collected and documented during the course of the study. For a period of 30 days following the last study drug administration, adverse events will also be documented if reported.
  Assessment of safety and tolerability to EP-7041, administered as a continuous IV infusion over 5 days, will be based on adverse events. Each AE will be graded with respect to its relationship to treatment using five categories: not related, unlikely, possible, probable, and highly probable. Each AE will also be graded on a 3-point severity scale: mild, moderate, and severe. Adverse events will be coded by body system and preferred term using the Medical Dictionary for Regulatory Activities dictionary. Assessments as to the effect of EP-7041 on vital signs, 12-lead ECG, telemetry, clinical laboratory parameters, physical examination, and local response to each injection, and body weight will also be made. The number and percentage of subjects experiencing adverse events will be tabulated for each treatment group by body system and preferred term.
  The number and percentage of subjects experiencing AEs will also be tabulated by relationship to drug treatment and by severity.

SECONDARY OUTCOMES:
Measurement of Maximum Plasma Concentration Achieved Following a Single IV Bolus of EP-7041 | 24 hours
  Maximum Plasma Concentration (Cmax)
Measurement of Time of Maximum Plasma Concentration Following a Single IV Bolus of EP-7041 | 24 hours
  Time of Maximum Plasma Concentration (Tmax)
Measurement of Plasma Half-Life Following a Single IV Bolus of EP-7041 | 24 hours
  Plasma Half-Life (T½)
Measurement of ClearanceFollowing a Single IV Bolus of EP-7041 | 24 hours
  Clearance (CL)
Measurement of the Area Under the Plasma Concentration versus Time Curve Following a Single IV Bolus of EP-7041 | 24 hours
  Area Under the Curve (AUC)
Measurement of the Elimination Rate Constant Following a Single IV Bolus of EP-7041 | 24 hours
  Elimination Rate Constant (Kel)
Measurement of the Apparent Volume of Distribution Following a Single IV Bolus of EP-7041 | 24 hours
  Apparent Volume of Distribution (Vd)
Measurement of the Steady-State Concentration with a the Initiation of Continuous IV 5-day Infusion of EP-7041 | 6 days
  Concentration at Steady State (Css)
Measurement of the Time to Reach a Steady-State Concentration Following a the Initiation of Continuous IV 5-day Infusion of EP-7041 | 6 days
  Time to Reach Concentration at Steady State (Tss)
Measurement of the Clearance During the Course of a Continuous IV 5-day Infusion of EP-7041 | 6 days
  Clearance (CL)
Measurement of the Plasma Half-Life Following the Discontinuation of Continuous IV 5-day Infusion of EP-7041 | 6 day
  Plasma Half-Life (T½)
Measurement of Clotting Biomarker Activated Partial Thromboplastin Time Following a Single IV Bolus of EP-7041 | 1 day
  Activated Partial Thromboplastin Time (aPTT)
Measurement of Clotting Biomarker Activated Partial Thromboplastin Time During the Course of a Continuous IV 5-day Infusion of EP-7041 | 6 days
  Activated Partial Thromboplastin Time (aPTT)
Measurement of Clotting Biomarker Prothrombin Following a Single IV Bolus of EP-7041 | 1 day
  Prothrombin Time (PT)
Measurement of Clotting Biomarker Prothrombin During the Course of a Continuous IV 5-day Infusion of EP-7041 | 6 day
  Prothrombin Time (PT)
Measurement of Clotting Biomarker International Normalized Ratio Following a Single IV Bolus of EP-7041 | 1 day
  International Normalized Ratio (INR)
Measurement of Clotting Biomarker International Normalized Ratio During the Course of a Continuous IV 5-day Infusion of EP-7041 | 6 days
  International Normalized Ratio (INR)

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — IDT CMAX
Locations (1):
- IDT CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No